CLINICAL TRIAL: NCT00706849
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Assess Efficacy and Safety of ISIS 301012 as Add-on Therapy in Heterozygous Familial Hypercholesterolemia Subjects With Coronary Artery Disease
Brief Title: Efficacy and Safety Study of ISIS 301012 (Mipomersen) as Add-on in Familial Hypercholesterolemic Patients With Coronary Artery Disease
Acronym: RADICHOL II
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kastle Therapeutics, LLC (Industry)
Collaborators: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 301012-CS7
Record Dates: First submitted 2008-06-26; First posted 2008-06-30 (Estimated); Results first posted 2013-03-21 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-08

CONDITIONS: Heterozygous Familial Hypercholesterolemia; Coronary Artery Disease
Keywords: familial hypercholesterolemia
MeSH Terms: conditions — Coronary Artery Disease; Hyperlipoproteinemia Type II | interventions — mipomersen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mipomersen (Experimental): Participants received mipomersen 200 mg as a subcutaneous injection once a week for 26 weeks.
  Interventions: Drug: mipomersen sodium
- Placebo (Placebo Comparator): Participants received a placebo subcutaneous injection once a week for 26 weeks.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: mipomersen sodium — 200 mg /mL
  Other Names: ISIS 301012; Kynamro™
  Arms: Mipomersen
Drug: placebo — 1 mL matching placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether mipomersen safely and effectively lowers low-density lipoprotein cholesterol (LDL-C) in patients with Heterozygous Familial Hypercholesterolemia (HeFH) and coronary artery disease (CAD) who are already on a stable dose of other lipid-lowering agents (including maximally tolerated statin therapy).

DETAILED DESCRIPTION:
Familial hypercholesterolemia (FH) is an autosomal dominant genetic disorder of lipoprotein metabolism characterized by markedly elevated LDL-C, premature onset of atherosclerosis and development of xanthomata. Patients with heterozygous familial hypercholesterolemia typically have total plasma cholesterol between 350 to 550 mg/dL and disease onset in their third and fourth decade.

Mipomersen (ISIS 301012) is an antisense drug that reduces a protein in the liver cells called apolipoprotein B (apo-B). Apo-B plays a role in producing low density lipoprotein cholesterol (the "bad" cholesterol) and moving it from the liver to one's bloodstream. High LDL-C is an independent risk factor for the development of coronary heart disease (CHD) or other diseases of blood vessels. It has been shown that lowering LDL-C reduces the risk of heart attacks and other major adverse cardiovascular events.

This study consisted of a 26-week treatment period and a 24-week post-treatment follow-up period (with the exception of patients who enrolled in the open-label extension study [Study 301012-CS6; NCT00694109]). The treatment period spanned the time during which the study treatment was administered until the later of the primary efficacy time point (PET) or 14 days beyond the last day of study drug administration. The post-treatment follow-up period began the day after completion of the treatment period and ended on the day of the patient's last contact date within the study.

Following treatment and Week 28 evaluations, eligible patients who tolerated study drug could elect to enroll in an open-label extension study (301012-CS6). Patients who were not eligible for or who elected not to enroll in the open-label extension study and patients who discontinued during the 26-week treatment period were followed in this study for an additional 24 weeks from administration of the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Heterozygous Familial Hypercholesterolemia (HeFH)
* Diagnosis of Coronary Artery Disease (CAD)
* Stable lipid-lowering therapy for 12 weeks
* On maximally tolerated statin therapy with at least 1 statin at a dose greater than zero, per Investigator judgment
* Stable low-fat diet for 8 weeks
* Stable weight for 6 weeks

Exclusion Criteria:

* Significant health problems in recent past including heart attack, stroke, coronary syndrome, unstable angina, heart failure, significant arrhythmia, orthostatic hypotension, uncontrolled hypertension, blood disorders, liver disease, cancer, or digestive problems
* Receiving apheresis treatment or last apheresis treatment within 8 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2008-07; Primary Completion 2009-12 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (44):
- United States (35):
  - La Jolla, California
  - Los Angeles, California
  - Mission Viejo, California
  - Newport Beach, California
  - Santa Ana, California
  - Thousand Oaks, California
  - Bridgeport, Connecticut
  - Melbourne, Florida
  - Pensacola, Florida
  - Chicago, Illinois
  - Naperville, Illinois
  - Kansas City, Kansas
  - Biddeford, Maine
  - Scarborough, Maine
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - St Louis, Missouri
  - Las Vegas, Nevada
  - Concord, New Hampshire
  - New York, New York
  - The Rogosin Institute Comprehensive Lipid Control Center, New York, New York
  - Charlotte, North Carolina
  - Durham, North Carolina
  - Cincinnati, Ohio
  - ResEvo, LLC, Cuyahoga Falls, Ohio
  - Franklin, Ohio
  - Oklahoma City, Oklahoma
  - Portland, Oregon
  - Nashville, Tennessee
  - Dallas, Texas
  - Grapevine, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Seattle, Washington
- Canada (9):
  - Calgary, Alberta
  - Vancouver, British Columbia
  - Winnipeg, Manitoba
  - London, Ontario
  - Toronto, Ontario
  - Chicoutimi, Quebec
  - Montreal, Quebec
  - Saint Foy, Quebec
  - Sherbrooke, Quebec

REFERENCES:
- [Result] Stein EA, Dufour R, Gagne C, Gaudet D, East C, Donovan JM, Chin W, Tribble DL, McGowan M. Apolipoprotein B synthesis inhibition with mipomersen in heterozygous familial hypercholesterolemia: results of a randomized, double-blind, placebo-controlled trial to assess efficacy and safety as add-on therapy in patients with coronary artery disease. Circulation. 2012 Nov 6;126(19):2283-92. doi: 10.1161/CIRCULATIONAHA.112.104125. Epub 2012 Oct 11. PMID 23060426
- [Derived] Duell PB, Santos RD, Kirwan BA, Witztum JL, Tsimikas S, Kastelein JJP. Long-term mipomersen treatment is associated with a reduction in cardiovascular events in patients with familial hypercholesterolemia. J Clin Lipidol. 2016 Jul-Aug;10(4):1011-1021. doi: 10.1016/j.jacl.2016.04.013. Epub 2016 May 9. PMID 27578134
- [Derived] Santos RD, Raal FJ, Catapano AL, Witztum JL, Steinhagen-Thiessen E, Tsimikas S. Mipomersen, an antisense oligonucleotide to apolipoprotein B-100, reduces lipoprotein(a) in various populations with hypercholesterolemia: results of 4 phase III trials. Arterioscler Thromb Vasc Biol. 2015 Mar;35(3):689-99. doi: 10.1161/ATVBAHA.114.304549. Epub 2015 Jan 22. PMID 25614280

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two hundred and twenty-five patients were screened and 124 participants were randomized on Day 1 in a 2:1 ratio to receive mipomersen or placebo once a week for 26 weeks.
Period: Treatment Period
Arm/Group | Placebo | Mipomersen
Started | 41 | 83
Full Analysis Set | 41 (Treated patients with a valid baseline & post-baseline LDL-C measurement) | 82 (Treated patients with a valid baseline & post-baseline LDL-C measurement.)
Completed | 41 (38 patients entered the open-label extension study (301012-CS6; NCT00694109).) | 73 (55 patients entered the open-label extension study (301012-CS6; NCT00694109).)
Not Completed | 0 | 10
Not completed — Adverse Event | 0 | 9
Not completed — Other | 0 | 1
Period: Follow-up Period
Arm/Group | Placebo | Mipomersen
Started | 3 (Participants enrolled in the open-label extension (NCT00694109) or continued in the follow-up period) | 28 (Participants enrolled in the open-label extension (NCT00694109) or continued in the follow-up period)
Completed | 3 | 25
Not Completed | 0 | 3
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Protocol non-compliance | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Mipomersen | Total
Number analyzed (Participants) | 41 | 83 | 124
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.9 (9.3) | 56.2 (9.7) | 56.1 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 33 | 46
  Male | 28 | 50 | 78
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 39 | 81 | 120
Race/Ethnicity, Customized [Number; unit: participants]
  White | 38 | 81 | 119
  Black | 1 | 2 | 3
  Other race | 2 | 0 | 2
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 30.25 (3.79) | 28.66 (4.23) | 29.18 (4.14)
Waist/hip ratio [Mean (Standard Deviation); unit: ratio] | 0.95 (0.07) | 0.93 (0.08) | 0.93 (0.08)
Metabolic syndrome [Number; unit: participants] — A patient was classified as having metabolic syndrome if any 3 of the following risk factors existed: 1) Waist circumference ≥102 cm (men) or ≥88 cm (women); 2) Triglycerides ≥150 mg/dl *; 3) High density lipoprotein cholesterol <40 mg/dl (men) or <50 mg/dl (women)*; 4) Systolic blood pressure ≥130 or diastolic ≥85 mmHg *; 5) Fasting glucose ≥100 mg/dl *.
  * = or on medication for the specified risk factor.
  participants
    No | 30 | 48 | 78
    Yes | 11 | 35 | 46
Tobacco use [Number; unit: participants]
  Current | 4 | 13 | 17
  non-current | 17 | 32 | 49
  Never | 20 | 38 | 58
Alcohol use [Number; unit: participants]
  Current | 31 | 64 | 95
  Non-current | 7 | 10 | 17
  Never | 3 | 9 | 12

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Low-density Lipoprotein Cholesterol (LDL-C) at the Primary Efficacy Time Point
Description: LDL cholesterol was measured in mg/dL. Samples were taken following an overnight fast. For patients with triglycerides <400 mg/dL, LDL-C was obtained using Friedewald's calculation; and for patients with triglycerides ≥400 mg/dL, LDL-C was directly measured by the central laboratory using ultracentrifugation. The primary efficacy time point was the post-baseline visit closest to 14 days after the last dose of study treatment.
Time Frame: Baseline (the average of the screening and Day 1 pre-treatment assessments) and the Primary Efficacy Time point (PET; Week 28 or the post-baseline visit closest to 14 days after the last dose).
Population: The Full Analysis Set, which consisted of all randomized patients who received at least 1 injection of study drug (mipomersen or placebo) and with a valid baseline and at least 1 post-baseline LDL-C measurement.
Measure: Mean (Standard Deviation); unit: percentage of Baseline
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 41 | 82
percentage of Baseline | 5.17 (18.02) | -28.02 (26.99)
Statistical Analysis 1: Comparison: Placebo vs Mipomersen; Based upon prior clinical study experience with mipomersen, it was estimated that the standard deviation of the percent change in LDL-C is approximately 22%. With 20 patients in the control group and 40 patients in the mipomersen-treated group, this study would have at least 90% power to detect a 20% difference between the 2 treatment groups; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — Statistical significance was concluded if p ≤ 0.05

2. Primary Outcome: LDL Cholesterol at Baseline and at the Primary Efficacy Time Point
Description: The primary efficacy time point (PET) was the post-baseline visit closest to 14 days after the last dose of study treatment.
Time Frame: as for outcome 1
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 41 | 82
mg/dL
  Baseline | 142.9 (51.6) | 152.9 (48.7)
  Primary efficacy time point | 146.4 (43.4) | 103.9 (33.0)

3. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B at the Primary Efficacy Time Point
Description: Apolipoprotein B was measured in mg/dL. Samples were taken following an overnight fast. The primary efficacy time point was the post-baseline visit closest to 14 days after the last dose of study treatment.
Time Frame: as for outcome 1
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: percentage of baseline
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 41 | 82
percentage of baseline | 7.02 (16.52) | -26.31 (22.16)
Statistical Analysis 1: Comparison: Placebo vs Mipomersen; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — Inflation of type 1 error was controlled by specifying a small number of secondary parameters and a sequential inferential approach in which inferential conclusions about each successive parameter required statistical significance of the prior one

4. Secondary Outcome: Apolipoprotein B at Baseline and at the Primary Efficacy Time Point
Description: as for outcome 2
Time Frame: as for outcome 1
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 41 | 82
mg/dL
  Baseline | 126.8 (33.2) | 132.8 (33.9)
  Primary efficacy time point | 133.8 (32.6) | 95.0 (29.7)

5. Secondary Outcome: Percent Change From Baseline in Total Cholesterol at the Primary Efficacy Time Point
Description: Total cholesterol was measured in mg/dL. Samples were taken following an overnight fast. The primary efficacy time point was the post-baseline visit closest to 14 days after the last dose of study treatment.
Time Frame: as for outcome 1
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: percentage of baseline
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 41 | 82
percentage of baseline | 3.85 (12.84) | -19.43 (19.25)
Statistical Analysis 1: Comparison: Placebo vs Mipomersen; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]

6. Secondary Outcome: Total Cholesterol at Baseline and at the Primary Efficacy Time Point
Description: as for outcome 2
Time Frame: as for outcome 1
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 41 | 82
mg/dL
  Baseline | 213.4 (54.6) | 225.3 (51.5)
  Primary efficacy time point | 219.0 (49.0) | 176.0 (35.9)

7. Secondary Outcome: Percent Change From Baseline in Non-High-Density Lipoprotein Cholesterol at the Primary Efficacy Time Point
Description: Non-high-density lipoprotein cholesterol was measured in mg/dL. Samples were taken following an overnight fast. The primary efficacy time point was the post-baseline visit closest to 14 days after the last dose of study treatment.
Time Frame: as for outcome 1
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: percentage of baseline
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 41 | 82
percentage of baseline | 3.74 (16.04) | -25.05 (25.71)
Statistical Analysis 1: Comparison: Placebo vs Mipomersen; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]

8. Secondary Outcome: Non-High-Density Lipoprotein Cholesterol at Baseline and at the Primary Efficacy Time Point
Description: as for outcome 2
Time Frame: as for outcome 1
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 41 | 82
mg/dL
  Baseline | 165.3 (54.5) | 175.5 (51.1)
  Primary efficacy time point | 168.2 (47.5) | 125.2 (37.8)

9. Other Pre Specified Outcome: Percent Change From Baseline in Triglycerides at the Primary Efficacy Time Point
Description: Triglycerides were measured in mg/dL. Samples were taken following an overnight fast. The primary efficacy time point was the post-baseline visit closest to 14 days after the last dose of study treatment.
Time Frame: as for outcome 1
Population: Full Analysis Set
Measure: Median (Inter-Quartile Range); unit: percentage of baseline
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 41 | 82
percentage of baseline | 0.5 (20.77) [-16.2 to 17.9] | -14.3 (43.76) [-32.7 to 9.7]
Statistical Analysis 1: Comparison: Placebo vs Mipomersen; Test type: Superiority or Other; p = 0.042, Wilcoxon (Mann-Whitney) — No adjustments were made for tertiary parameters

10. Other Pre Specified Outcome: Triglycerides at Baseline and at the Primary Efficacy Time Point
Description: as for outcome 2
Time Frame: as for outcome 1
Population: Full Analysis Set
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 41 | 82
mg/dL
  Baseline | 100 (53.3) [74 to 137] | 107 (39.6) [85 to 137]
  Primary efficacy time point | 101 (42.5) [76 to 139] | 89 (70.1) [70 to 127]

11. Other Pre Specified Outcome: Percent Change From Baseline in Lipoprotein (a) at the Primary Efficacy Time Point
Description: Lipoprotein (a) was measured in mg/dL. Samples were taken following an overnight fast. The primary efficacy time point was the post-baseline visit closest to 14 days after the last dose of study treatment.
Time Frame: as for outcome 1
Population: Full Analysis Set
Measure: Median (Inter-Quartile Range); unit: percentage of baseline
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 41 | 82
percentage of baseline | 0.0 (15.10) [-8.0 to 13.0] | -21.1 (24.22) [-37.9 to 0.0]
Statistical Analysis 1: Comparison: Placebo vs Mipomersen; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — No adjustments were made for tertiary parameters

12. Other Pre Specified Outcome: Lipoprotein (a) at Baseline and at the Primary Efficacy Time Point
Description: as for outcome 2
Time Frame: as for outcome 1
Population: Full Analysis Set
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 41 | 82
mg/dL
  Baseline | 53 (56.2) [17 to 108] | 45 (64.6) [13 to 93]
  Primary efficacy time point | 51 (53.5) [18 to 108] | 35 (55.3) [9 to 56]

13. Other Pre Specified Outcome: Percent Change From Baseline in Very Low Density Lipoprotein Cholesterol at the Primary Efficacy Time Point
Description: Very low density lipoprotein (VLDL) cholesterol was measured in mg/dL. Samples were taken following an overnight fast. The primary efficacy time point was the post-baseline visit closest to 14 days after the last dose of study treatment.
Time Frame: as for outcome 1
Population: Full Analysis Set
Measure: Median (Inter-Quartile Range); unit: percentage of baseline
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 41 | 82
percentage of baseline | 0.0 (20.11) [-15.4 to 15.0] | -13.8 (45.70) [-33.3 to 11.8]
Statistical Analysis 1: Comparison: Placebo vs Mipomersen; Test type: Superiority or Other; p = 0.023, Wilcoxon (Mann-Whitney) — No adjustments were made for tertiary parameters

14. Other Pre Specified Outcome: Very Low Density Lipoprotein at Baseline and at the Primary Efficacy Time Point
Description: as for outcome 2
Time Frame: as for outcome 1
Population: Full Analysis Set
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 41 | 82
mg/dL
  Baseline | 20 (9.5) [15 to 28] | 21 (7.9) [17 to 27]
  Primary efficacy time point | 20 (8.5) [15 to 28] | 18 (14.6) [14 to 25]

15. Other Pre Specified Outcome: Percent Change From Baseline in the Ratio of LDL Cholesterol to HDL Cholesterol at the Primary Efficacy Time Point
Description: The ratio of low-density lipoprotein (LDL) cholesterol to high-density lipoprotein (HDL) cholesterol was measured at Baseline and the post-baseline visit closest to 14 days after the last dose of study treatment.
Time Frame: as for outcome 1
Population: Full Analysis Set
Measure: Median (Inter-Quartile Range); unit: percentage of baseline
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 41 | 82
percentage of baseline | -2.8 (19.38) [-13.1 to 13.1] | -29.2 (29.99) [-46.8 to -13.7]
Statistical Analysis 1: Comparison: Placebo vs Mipomersen; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — No adjustments were made for tertiary parameters

16. Other Pre Specified Outcome: Ratio of LDL Cholesterol to HDL Cholesterol at Baseline and at the Primary Efficacy Time Point
Description: as for outcome 2
Time Frame: as for outcome 1
Population: Full Analysis Set
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 41 | 82
ratio
  Baseline | 2.72 (1.495) [2.51 to 3.34] | 2.99 (1.353) [2.56 to 4.00]
  Primary efficacy time point | 2.95 (1.337) [2.19 to 3.49] | 2.09 (1.034) [1.52 to 3.00]

17. Other Pre Specified Outcome: Percent Change From Baseline in Apolipoprotein A1 at the Primary Efficacy Time Point
Description: Apolipoprotein A1 was measured in mg/dL. Samples were taken following an overnight fast. The primary efficacy time point was the post-baseline visit closest to 14 days after the last dose of study treatment.
Time Frame: as for outcome 1
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: percentage of baseline
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 41 | 82
percentage of baseline | 3.71 (8.70) | -2.44 (14.22)
Statistical Analysis 1: Comparison: Placebo vs Mipomersen; Test type: Superiority or Other; p = 0.004, t-test, 2 sided — No adjustments were made for tertiary parameters

18. Other Pre Specified Outcome: Apolipoprotein A1 at Baseline and at the Primary Efficacy Time Point
Description: as for outcome 2
Time Frame: as for outcome 1
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 41 | 82
mg/dL
  Baseline | 146.1 (24.9) | 150.7 (28.1)
  Primary efficacy time point | 151.5 (29.1) | 145.4 (27.9)

19. Other Pre Specified Outcome: Percent Change From Baseline in High-Density Lipoprotein Cholesterol at the Primary Efficacy Time Point
Description: High-density lipoprotein cholesterol (HDL-C) was measured in mg/dL. Samples were taken following an overnight fast. The primary efficacy time point was the post-baseline visit closest to 14 days after the last dose of study treatment.
Time Frame: as for outcome 1
Population: Full Analysis Set
Measure: Median (Inter-Quartile Range); unit: percentage of baseline
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 41 | 82
percentage of baseline | 5.8 (9.57) [0.0 to 11.5] | 2.5 (18.04) [-10.3 to 11.7]
Statistical Analysis 1: Comparison: Placebo vs Mipomersen; Test type: Superiority or Other; p = 0.207, Wilcoxon (Mann-Whitney) — No adjustments were made for tertiary parameters

20. Other Pre Specified Outcome: High-Density Lipoprotein Cholesterol at Baseline and at the Primary Efficacy Time Point
Description: as for outcome 2
Time Frame: as for outcome 1
Population: Full Analysis Set
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 41 | 82
mg/dL
  Baseline | 48 (11.1) [41 to 53] | 47 (13.6) [40 to 58]
  Primary efficacy time point | 51 (13.5) [42 to 58] | 48 (15.6) [40 to 58]

ADVERSE EVENTS:
Time Frame: Up to Week 28 (2 weeks after last dose)
Description: In the event a single participant has experienced both a serious and a non-serious form of the same adverse event term, the individual has been included in the numerator ("number of affected participants") of both adverse event tables.
Arm/Group | Placebo | Mipomersen
Serious Adverse Events (participants affected / at risk) | 2/41 | 6/83
Other Adverse Events (participants affected / at risk) | 38/41 | 83/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=41) | Mipomersen (N=83)
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Chest pain (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=41) | Mipomersen (N=83)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 1
Angina pectoris (Cardiac disorders) | 0 | 2
Coronary artery disease (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 1
Palpitations (Cardiac disorders) | 0 | 2
Sinus bradycardia (Cardiac disorders) | 1 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 1
Cataract (Eye disorders) | 0 | 1
Conjunctivitis (Eye disorders) | 0 | 1
Dry eye (Eye disorders) | 0 | 1
Eye irritation (Eye disorders) | 0 | 1
Eyelid cyst (Eye disorders) | 0 | 1
Presbyopia (Eye disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 2
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 6
Bezoar (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 3 | 4
Dental caries (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 9
Diverticulum (Gastrointestinal disorders) | 1 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 3
Dysphagia (Gastrointestinal disorders) | 0 | 1
Gastric polyps (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Haematochezia (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 1
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 1 | 0
Lip pain (Gastrointestinal disorders) | 0 | 1
Lip swelling (Gastrointestinal disorders) | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 6 | 14
Oesophageal dilatation (Gastrointestinal disorders) | 0 | 1
Paraesthesia oral (Gastrointestinal disorders) | 0 | 1
Periodontal disease (Gastrointestinal disorders) | 0 | 1
Retching (Gastrointestinal disorders) | 0 | 1
Tooth disorder (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 5
Adverse drug reaction (General disorders) | 0 | 1
Asthenia (General disorders) | 2 | 1
Chills (General disorders) | 1 | 6
Cyst (General disorders) | 1 | 0
Discomfort (General disorders) | 1 | 1
Facial pain (General disorders) | 0 | 1
Fatigue (General disorders) | 4 | 22
Feeling jittery (General disorders) | 0 | 1
Influenza like illness (General disorders) | 3 | 15
Injection site discolouration (General disorders) | 1 | 13
Injection site discomfort (General disorders) | 0 | 10
Injection site eczema (General disorders) | 0 | 1
Injection site erythema (General disorders) | 3 | 56
Injection site haematoma (General disorders) | 9 | 45
Injection site haemorrhage (General disorders) | 1 | 9
Injection site induration (General disorders) | 0 | 11
Injection site inflammation (General disorders) | 0 | 3
Injection site lymphadenopathy (General disorders) | 0 | 1
Injection site macule (General disorders) | 0 | 3
Injection site nodule (General disorders) | 0 | 8
Injection site oedema (General disorders) | 0 | 6
Injection site pain (General disorders) | 8 | 54
Injection site papule (General disorders) | 0 | 5
Injection site paraesthesia (General disorders) | 0 | 2
Injection site pruritus (General disorders) | 2 | 23
Injection site rash (General disorders) | 0 | 11
Injection site reaction (General disorders) | 1 | 5
Injection site recall reaction (General disorders) | 0 | 15
Injection site swelling (General disorders) | 0 | 13
Injection site urticaria (General disorders) | 0 | 3
Injection site vesicles (General disorders) | 0 | 2
Injection site warmth (General disorders) | 0 | 12
Injury associated with device (General disorders) | 0 | 1
Irritability (General disorders) | 0 | 2
Local swelling (General disorders) | 0 | 1
Localised oedema (General disorders) | 0 | 1
Malaise (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 2
Oedema peripheral (General disorders) | 1 | 7
Pain (General disorders) | 3 | 5
Pyrexia (General disorders) | 0 | 10
Tenderness (General disorders) | 0 | 1
Vessel puncture site haematoma (General disorders) | 0 | 1
Hepatic cyst (Hepatobiliary disorders) | 0 | 1
Hepatic lesion (Hepatobiliary disorders) | 1 | 0
Hepatic steatosis (Hepatobiliary disorders) | 0 | 5
Hepatomegaly (Hepatobiliary disorders) | 0 | 1
Abscess oral (Infections and infestations) | 1 | 0
Asymptomatic bacteriuria (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0
Ear infection (Infections and infestations) | 1 | 0
Eye infection (Infections and infestations) | 1 | 0
Eye infection viral (Infections and infestations) | 1 | 0
Furuncle (Infections and infestations) | 1 | 0
Gastrointestinal infection (Infections and infestations) | 1 | 0
Gastrointestinal viral infection (Infections and infestations) | 0 | 2
H1N1 influenza (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 2 | 5
Kidney infection (Infections and infestations) | 0 | 2
Laryngitis (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Lyme disease (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 3 | 9
Pneumonia (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 0
Rhinitis (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 4 | 1
Upper respiratory tract infection (Infections and infestations) | 3 | 4
Urinary tract infection (Infections and infestations) | 4 | 6
Vaginal infection (Infections and infestations) | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 0
Animal bite (Injury, poisoning and procedural complications) | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 1 | 0
Brain contusion (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 5
Epicondylitis (Injury, poisoning and procedural complications) | 0 | 1
Face injury (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Injury (Injury, poisoning and procedural complications) | 0 | 1
Joint sprain (Injury, poisoning and procedural complications) | 1 | 0
Muscle injury (Injury, poisoning and procedural complications) | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 1 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Scratch (Injury, poisoning and procedural complications) | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0
Sunburn (Injury, poisoning and procedural complications) | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 6
Aspartate aminotransferase increased (Investigations) | 1 | 3
Bacterial test positive (Investigations) | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 2 | 0
Blood pressure increased (Investigations) | 1 | 0
Body temperature increased (Investigations) | 0 | 2
Carotid bruit (Investigations) | 1 | 1
Computerised tomogram abdomen abnormal (Investigations) | 0 | 1
Electrocardiogram T wave inversion (Investigations) | 0 | 1
Epstein-Barr virus antibody positive (Investigations) | 0 | 1
Haematocrit decreased (Investigations) | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 4
Herpes simplex serology positive (Investigations) | 0 | 1
International normalised ratio increased (Investigations) | 0 | 2
Liver function test abnormal (Investigations) | 1 | 5
Multiple gated acquisition scan abnormal (Investigations) | 0 | 1
Nitrite urine present (Investigations) | 0 | 1
Nuclear magnetic resonance imaging abnormal (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 0 | 2
Protein urine present (Investigations) | 0 | 1
Pulse abnormal (Investigations) | 0 | 1
Red blood cells urine positive (Investigations) | 0 | 1
Transaminases increased (Investigations) | 0 | 2
Urine leukocyte esterase positive (Investigations) | 0 | 1
Weight decreased (Investigations) | 1 | 1
Weight increased (Investigations) | 1 | 1
White blood cells urine positive (Investigations) | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 3 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 6
Axillary mass (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 7
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint warmth (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 8
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 4
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spondylitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Morton's neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Amnesia (Nervous system disorders) | 1 | 0
Burning sensation (Nervous system disorders) | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 1 | 0
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0
Disturbance in attention (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 4 | 4
Dizziness postural (Nervous system disorders) | 0 | 2
Dysgeusia (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 7 | 15
Hyperaesthesia (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 0 | 2
Migraine with aura (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 4
Sciatica (Nervous system disorders) | 0 | 2
Sinus headache (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 2 | 3
Claustrophobia (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 2
Libido decreased (Psychiatric disorders) | 0 | 1
Panic attack (Psychiatric disorders) | 0 | 1
Stress (Psychiatric disorders) | 0 | 1
Albuminuria (Renal and urinary disorders) | 0 | 1
Chromaturia (Renal and urinary disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Micturition urgency (Renal and urinary disorders) | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 2
Proteinuria (Renal and urinary disorders) | 0 | 3
Stress urinary incontinence (Renal and urinary disorders) | 0 | 1
Urge incontinence (Renal and urinary disorders) | 0 | 1
Menstruation delayed (Reproductive system and breast disorders) | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 0
Prostatomegaly (Reproductive system and breast disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 7
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 2
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 1
Hypoaesthesia facial (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 2
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 4 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Scab (Skin and subcutaneous tissue disorders) | 0 | 1
Skin induration (Skin and subcutaneous tissue disorders) | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0
Skin plaque (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Aortic aneurysm (Vascular disorders) | 0 | 1
Flushing (Vascular disorders) | 1 | 1
Hot flush (Vascular disorders) | 0 | 3
Hypertension (Vascular disorders) | 1 | 2
Hypotension (Vascular disorders) | 0 | 1
Infarction (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After the multicenter publication or 12 months after completion of the study the PI may publish the results of his/her data from the study. The PI shall provide the sponsor with an advance copy at least 60 days prior to planned submission and the Sponsor shall have 60 days to review (contracts have variable timeframes; maximum times are stated here). The sponsor may request the deletion of any confidential information, or a delay in submission for an additional period not to exceed 90 days.